CLINICAL TRIAL: NCT04970004
Title: A Retrospective Observational Study of Adult and Pediatric Patients With Thrombotic Microangiopathy (TMA) After Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: Study in Adult and Pediatric Patients With HSCT-TMA
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision to not proceed.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALX-TMA-501
Record Dates: First submitted 2021-07-16; First posted 2021-07-21 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Stem Cell Transplant Complications; Thrombotic Microangiopathies
Keywords: Hematopoietic Stem Cell Transplant; Transplant-associated TMA; Thrombotic Microangiopathy (TMA)
MeSH Terms: conditions — Thrombotic Microangiopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Diagnosed with HSCT-TMA
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No study intervention will be administered as part of this study.

SUMMARY:
This is an observational, retrospective study designed to assess outcomes in patients diagnosed with hematopoietic stem cell transplant-associated thrombotic microangiopathy (HSCT-TMA) who were not treated with complement component (C5) inhibitor therapy. Data required to evaluate study outcomes will be abstracted from the medical records of all patients who meet study eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 5 kg at the time of HSCT-TMA diagnosis
* Documented TMA diagnosis within 6 months from the HSCT
* Evidence of renal dysfunction
* Presence of hypertension

Exclusion Criteria:

* History or presence of familial or acquired 'a disintegrin and metalloproteinase with a thrombospondin type 1 motif, member 13' (ADAMTS13) deficiency (activity < 5%)
* Shiga toxin-related hemolytic uremic syndrome (ST-HUS)
* Positive direct Coombs test
* Diagnosis of disseminated intravascular coagulation
* History or presence of bone marrow/graft failure
* Diagnosis of veno-occlusive disease
* Received a complement inhibitor (eg, eculizumab) post-HSCT through 12 months post TMA diagnosis

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients who were diagnosed with TMA within 6 months after a HSCT procedure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving TMA Response | During the 26-week period after HSCT-TMA diagnosis
  TMA Response is defined as platelet count ≥ 50,000/mm^3, lactate dehydrogenase < 1.5 upper limit of normal, absence of schistocytes (if present at baseline), and increase in eGFR ≥ 30% from baseline or discontinuation of dialysis (for patients on dialysis at baseline)

SECONDARY OUTCOMES:
Proportion of patients achieving TMA response | During the 52-week period after HSCT-TMA diagnosis
Changes in individual components of TMA response | From baseline to 26 weeks and to 52 weeks after HSCT-TMA diagnosis
  Platelets, lactate dehydrogenase, eGFR, chronic kidney disease stage, dialysis status
Overall survival | At 26 weeks and 52 weeks after HSCT-TMA diagnosis
Nonrelapse mortality | At 26 weeks and 52 weeks after HSCT-TMA diagnosis
  Death due to any cause during the study, with the exception of death due to underlying disease progression or relapse

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No